CLINICAL TRIAL: NCT05519865
Title: A Randomized, Double-blind, Controlled, Multi-center Phase II Clinical Trial of Tucidinostat Combined With Tislelizumab as First-line Treatment for PD-L1 Positive Locally Advanced or Metastatic Non-Small Cell Lung Cancer
Brief Title: A Study of Tucidinostat Combined With Tislelizumab as First-line Treatment in Advanced NSCLC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chipscreen Biosciences, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CDM206
Record Dates: First submitted 2022-08-23; First posted 2022-08-29 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; tislelizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tucidinostat Combined with Tislelizumab (Experimental): Subjects receive Tucidinostat 30mg orally biw and Tislelizumab 200 mg intravenously (IV) Q3W.
  Interventions: Drug: Tucidinostat; Drug: Tislelizumab
- Tislelizumab (Active Comparator): Subjects receive Tislelizumab 200 mg intravenously (IV) Q3W.
  Interventions: Drug: Tislelizumab

INTERVENTIONS:
Drug: Tucidinostat — 30mg orally BIW
  Other Names: Chidamide; CS055
  Arms: Tucidinostat Combined with Tislelizumab
Drug: Tislelizumab — 200 mg intravenously (IV) Q3W

SUMMARY:
A Randomized, Double-blind, Controlled, Multi-center Phase 2 Clinical study to Investigate the Efficacy and Safety of Tucidinostat (Chidamide) Combined with Tislelizumab as First-line Treatment for PD-L1 Positive Locally Advanced or Metastatic Non-Small Cell Lung Cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years, Male or female.
2. Histologically or cytologically confirmed diagnosis of unresectable locally advanced or metastatic (stage IIIB-IV) NSCLC.
3. Must have no prior systemic anti-tumor therapy for locally advanced or metastatic NSCLC.
4. Must have positive PD-L1 expression in tumor tissue.
5. ECOG performance status of 0 or 1.
6. Must Have ≥1 measurable target lesion as defined by RECIST v.1.1.
7. Must have adequate organ function.
8. Life expectancy ≥ 12 weeks.
9. Signed informed consent form (ICF).

Exclusion Criteria:

1. With EGFR or ALK gene mutation.
2. Received prior targeted therapy.
3. Prior use of HDAC inhibitor.
4. Received prior therapies targeting PD-1, PD-L1, CTLA4, or any other immune checkpoint pathway.
5. Received any anti-tumor therapy or investigational agent and device within 28 days before the first dose of study treatment.
6. Received radiotherapy within 2 weeks or thoracic radiation >30Gy within 6 months before the first dose of study treatment.
7. Received systemic immunosuppressive drugs within 28 days before the first dose of study treatment. Inhaled or topical steroids and physiological dose of systemic glucocorticoid (≤10 mg daily prednisone equivalents) are permitted.
8. Received systemic immunostimulatory drugs within 28 days before the first dose of study treatment.
9. Received a live vaccine within 28 days before the first dose of study treatment or planned to receive during the study period. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; and COVID-19 vaccine also are allowed.
10. Received major surgery within 28 days before the first dose of study treatment.
11. Has not recovered ( ≤ Grade 1 defined by CTCAE V5.0) from AEs due to prior anti-cancer therapy.
12. Has symptomatic and untreated central nervous system (CNS) metastases.
13. Has hydrothorax and ascites with obvious symptoms or requiring repeated drainage within 1 month before the first dose of study treatment.
14. Uncontrollable or major cardiovascular and cerebrovascular disease.
15. History of hemoptysis within 2 weeks or active bleeding within 2 months before the first dose of study treatment; or subject who is taking anticoagulants, or subject with clear high-risk bleeding tendency during the screening period.
16. History of serious thromboembolism within 6 months before the first dose of study treatment.
17. Suspected interstitial lung disease (ILD) or pulmonary fibrosis or pulmonary inflammation requiring treatment; or history of lung disease treated with oral or intravenous steroids within 6 months before the first dose of study treatment.
18. Obvious gastrointestinal abnormalities during the screening period, which may affect the intake, transport or absorption of drugs.
19. Urinary protein ≥ 2+ and quantitative urinary protein ≥ 1g/24 h during the screening period.
20. Active infection requiring intravenous therapy; or severe infection within 28 days before the first dose of study treatment.
21. Known active pulmonary tuberculosis, or subject who is receiving antituberculous treatment or having received antituberculous treatment within 1 year before the first dose of study treatment.
22. Active hepatitis B or hepatitis C.
23. HIV positive or history of AIDS or other serious infectious diseases.
24. History of malignant tumor.
25. Active autoimmune diseases during the screening period, and have received systemic treatment within 2 years before the first dose of study treatment.
26. History of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation.
27. Contraindications to any of the study drug ingredients.
28. History of hypersensitivity to monoclonal antibody, Chidamide, study drugs, or any of its excipients.
29. History of alcohol or drug abuse.
30. Unwilling or unable to comply with procedures required in this protocol.
31. Pregnant or breast-feeding women. Male/Female is unwilling or unable to use a highly effective method of birth control.

33. Any condition not suitable for participating in the trial in the opinion of the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2022-10-26 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) per RECIST v1.1 | Up to 2 years
  PFS assessed by investigator per RECIST v1.1, measured from the date of randomization until progression or death, whichever is first met.

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to 2 years
  Proportion of participants who have a partial response (PR) or complete response (CR) to therapy according to RECIST 1.1 or iRECIST.
Progression Free Survival (PFS) per iRECIST | Up to 2 years
  PFS assessed by investigator per iRECIST, measured from the date of randomization until progression or death, whichever is first met.
Overall Survival (OS) | Up to 2 years
  From the first dose of treatment until the date of death from any cause.
Disease control rate (DCR) | Up to 2 years
  Proportion of participants in partial, complete or stable disease according to RECIST 1.1 or iRECIST.
Duration of response (DOR) | Up to 2 years
  From the first date of response until the date of first documented progression according to RECIST 1.1 or iRECIST.
Progression-free survival of 6 months | 6 months after randomization
  Proportion of subjects who did not have disease progression(according to RECIST1.1 or iRECIST) or death at 6 months after randomization.
time to progression (TTP) | Up to 2 years
  TTP is measured from date of randomization until progression(according to RECIST1.1 or iRECIST) not including death.
time to response (TTR) | Up to 2 years
  TTR is measured from date of randomization until response
Safety and Tolerability | Up to 2 years
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Caicun Zhou, Principal Investigator — caicunzhoudr@163.com
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No